CLINICAL TRIAL: NCT06490744
Title: Evolution of Respiratory Function in Lung Transplant Patients With Moderate to Severe SARS-Cov-2 Infection, Single-center Retrospective Study
Brief Title: Evolution of Respiratory Function in Lung Transplant Patients With Moderate to Severe Covid-19 Infection
Acronym: Cov- EvoLuT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9058
Record Dates: First submitted 2024-07-04; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: COVID-19 Respiratory Infection
Keywords: Covid-19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; SARS-Cov-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SARS-Cov-2 infection pandemic has caused a large number of acute respiratory failures and deaths across the world. Certain factors have been identified as associated with a higher risk of developing a severe form and dying. Immunosuppression has been identified as a risk factor for progressing to a severe form.

Lung transplant patients were particularly vulnerable during this period, with a high frequency of respiratory compromise, sometimes progressing towards acute respiratory distress syndrome and, at a later stage, towards fibrotic forms. The impact of the infection on the immunological status of the patient and on the tolerance of the transplant have been little studied. The various treatments implemented during the pandemic have rapidly evolved (immunotherapy, vaccination, convalescent plasma transfusion, etc.) which may have modulated this risk. The evolution of respiratory function may be linked to the respiratory infection itself, or to the severity of respiratory damage during the infection. It is therefore relevant to compare patients with a moderate form of COVID-19 (non-intubated patients) to patients with severe forms, requiring invasive ventilation in intensive care. The evolution of respiratory function after infection has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Lung transplant patient (monopulmonary or bipulmonary)
* Covid diagnosed by RT-PCR between March 1, 2020 and December 31, 2022
* Hospitalization at the University Hospitals of Strasbourg for COVID-19
* Patient followed in the context of their lung transplant at the University Hospitals of Strasbourg
* Absence of written opposition in the subject's medical file to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed his opposition to the reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult lung transplant patients who had a Covid-19 infection and were treated at the Strasbourg University Hospital during the period from March 1, 2020 to December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the evolution of respiratory function in lung transplant recipients after moderate to severe Covid-19. | Files analyzed retrospectively cover the period from March 1, 2020 to December 31, 2022.
  This retrospective study concerns lung transplant patients who had a Covid-19 infection and were treated at the Strasbourg University Hospital during the period from March 1, 2020 to December 31, 2022.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation - CHU de Strasbourg - France, Strasbourg, France